CLINICAL TRIAL: NCT04324788
Title: Investigation of the Effect of Stair Activity on Lumbal Paravertebral Mechanical Properties in Transtibial and Transfemoral Amputes.
Brief Title: Investigation of the Effect of Stair Activity on Lumbal Paravertebral Mechanical Properties in Amputes.
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2019.969
Record Dates: First submitted 2020-03-24; First posted 2020-03-27 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Stair up and Down, Amputation; Amputation,Stair up and Down

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Transtibial amputation
  The patients will be asked to go up and down 9-step stair with the highest speed they can make.
  Interventions: Other: Group 1
- Group 2: Transfemoral amputation
  The patients will be asked to go up and down 9-step stair with the highest speed they can make.
  Interventions: Other: Group 2

INTERVENTIONS:
Other: Group 1 — The patients will be asked to go up and down 9-step stair with the highest speed they can make.
  Groups: Group 1
Other: Group 2 — The patients will be asked to go up and down 9-step stair with the highest speed they can make.
  Groups: Group 2

SUMMARY:
With the onset of prosthesis use following lower extremity amputations,body shows biomechanical changes according to the amputation level and consequently develops adaptation mechanisms both on the healthy and ampute side. Adaptations in the lumbo-pelvic and lower lumbar regions cause asymmetries in the muscle tissue by causing changes in the morphological structure of the muscle, especially in the muscles of the waist, hip and knee and recruitment.

The aim of this study is to investigate the effect of stairing up and down activity on the mechanical properties of lumbal paravertebral muscles in TFA and TTA and its relation with lower lumbar region pain.

ELIGIBILITY:
Inclusion Criteria:

* to be TTA and TFA
* No complaints of chronic low back pain before amputation
* Using prosthesis for at least 6 months
* Being able to climb up and down stairs
* No history of falls that will cause injury or pain in the past 6 months
* Having good prosthesis comfort
* BMI<28.5
* Who can have cognitive functions to understand Arabic language

Exclusion Criteria:

* To be amputated due to congenital and tumor
* Who can not have cognitive functions to understand Arabic language
* Having orthopedic or neurological disorders that may cause chronic pain or functional impairment in the lumbar region
* Ankylosing spondolitis and rheumatoid arthritis patients

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — with unilateral transtibial/transfemoral amputation
Study Population: Unilateral transfemoral and transtibial amputate patients
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Evaluation of the mechanical properties of the muscle-1 | Change from Baseline mechanical properties at following staring up and down activity, at 10 minutes after the staring up and down activity
  Viscoelastic stiffness [N/m] will be measured in MyotonPro 3 (MYO, Tallin, Estonia
Evaluation of the mechanical properties of the muscle-2 | Change from Baseline mechanical properties at following staring up and down activity, at 10 minutes after the staring up and down activity
  Oscillation frequency (Hz) will be measured in MyotonPro 3 (MYO, Tallin, Estonia
Evaluation of the mechanical properties of the muscle-3 | Change from Baseline mechanical properties at following staring up and down activity, at 10 minutes after the staring up and down activity
  Mechanical stiffness (N/m) will be measured in MyotonPro 3 (MYO, Tallin, Estonia
Evaluation of the back pain | Change from Baseline mechanical properties at following staring up and down activity, at 10 minutes after the staring up and down activity
  Pain will be evaluated by using Visual analog scale ranging 0 (no pain)- 10 (worst pain)
Evaluation of the pressure-pain threshold | Change from Baseline mechanical properties at following staring up and down activity, at 10 minutes after the staring up and down activity
  The pressure-pain threshold (lbs) will be measured in algometer commander (JTECH MEDICAL, MM036_K, 2016)

CONTACTS AND LOCATIONS:
Locations (1):
- Yasar Tatar, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Devan H, Hendrick P, Ribeiro DC, Hale LA, Carman A. Asymmetrical movements of the lumbopelvic region: is this a potential mechanism for low back pain in people with lower limb amputation? Med Hypotheses. 2014 Jan;82(1):77-85. doi: 10.1016/j.mehy.2013.11.012. Epub 2013 Nov 16. PMID 24296234
- [Background] Hendershot BD, Bazrgari B, Nussbaum MA. Persons with unilateral lower-limb amputation have altered and asymmetric trunk mechanical and neuromuscular behaviors estimated using multidirectional trunk perturbations. J Biomech. 2013 Jul 26;46(11):1907-12. doi: 10.1016/j.jbiomech.2013.04.018. Epub 2013 May 29. PMID 23726183
- [Background] Highsmith MJ, Kahle JT, Kaluf B, Miro RM, Mengelkoch LJ, Klenow TD. PSYCHOMETRIC EVALUATION OF THE HILL ASSESSMENT INDEX (HAI) AND STAIR ASSESSMENT INDEX (SAI) IN HIGH-FUNCTIONING TRANSFEMORAL AMPUTEES. Technol Innov. 2016 Sep;18(2-3):193-201. doi: 10.21300/18.2-3.2016.193. PMID 28066528
- [Background] Hu X, Lei D, Li L, Leng Y, Yu Q, Wei X, Lo WLA. Quantifying paraspinal muscle tone and stiffness in young adults with chronic low back pain: a reliability study. Sci Rep. 2018 Sep 25;8(1):14343. doi: 10.1038/s41598-018-32418-x. PMID 30254233
- [Background] Michaud SB, Gard SA, Childress DS. A preliminary investigation of pelvic obliquity patterns during gait in persons with transtibial and transfemoral amputation. J Rehabil Res Dev. 2000 Jan-Feb;37(1):1-10. PMID 10847567
- [Background] Kelly-Martin R, Doughty L, Garkavi M, Wasserman JB. Reliability of modified adheremeter and digital pressure algometer in measuring normal abdominal tissue and C-section scars. J Bodyw Mov Ther. 2018 Oct;22(4):972-979. doi: 10.1016/j.jbmt.2018.02.017. Epub 2018 Feb 17. PMID 30368344